CLINICAL TRIAL: NCT05402527
Title: Effects of a Nutritional Supplement of Proteins, ω3 Fatty Acids and Vitamin D on Physical Performance, Body Composition and Biochemical Profile of Persons Following High-intensity Functional Training
Brief Title: Fish Nutrient Supplementation in High-intensity Functional Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: AQUABIOPRO-FIT1
Record Dates: First submitted 2022-04-22; First posted 2022-06-02 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Exercise Training; Dietary Supplements
MeSH Terms: interventions — Whey Proteins; maltodextrin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are instructed not to disclose the supplement they are taking to their trainers, investigators, or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Fish nutrients - Whey protein - Maltodextrin (Other): Participants will receive fish nutrients, whey protein, and maltodextrin in this order.
  Interventions: Dietary Supplement: Fish nutrients; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Fish nutrients - Maltodextrin - Whey protein (Other): Participants will receive fish nutrients, maltodextrin, and whey protein in this order.
  Interventions: Dietary Supplement: Fish nutrients; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Whey protein - Fish nutrients - Maltodextrin (Other): Participants will receive whey protein, fish nutrients, and maltodextrin in this order.
  Interventions: Dietary Supplement: Fish nutrients; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Whey protein - Maltodextrin - Fish nutrients (Other): Participants will receive whey protein, maltodextrin, and fish nutrients in this order.
  Interventions: Dietary Supplement: Fish nutrients; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Maltodextrin - Fish nutrients - Whey protein (Other): Participants will receive maltodextrin, fish nutrients, and whey protein in this order.
  Interventions: Dietary Supplement: Fish nutrients; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin
- Maltodextrin - Whey protein - Fish nutrients (Other): Participants will receive maltodextrin, whey protein, and fish nutrients in this order.
  Interventions: Dietary Supplement: Fish nutrients; Dietary Supplement: Whey protein; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Fish nutrients — Intake of fish protein, omega-3 fatty acids, and vitamin D
Dietary Supplement: Whey protein — Intake of whey protein
Dietary Supplement: Maltodextrin — Intake of maltodextrin

SUMMARY:
Nowadays, many persons who exercise consume dietary supplements. Previous scientific studies have found that protein supplementation increases muscle mass when combined with an exercise program. In addition, vitamin D probably improves performance and muscle function. Likewise, ω3 fatty acids, apart from improving cardiovascular function, may also increase protein synthesis and performance. Thus, the aim of this study is to investigate the efficacy of a novel aquaculture-based sport supplement of proteins, ω3 fatty acids and vitamin D on physical performance, body composition, and the biochemical profile of persons following high-intensity functional training (HIFT). The efficacy of the experimental supplement (E) will be compared with whey protein (W) and maltodextrin (a carbohydrate) as placebo (P).

Thirty healthy trained individuals (15 male and 15 female), aged 18-35, will take E, W, and P during three 6-week periods of HIFT (a different supplement each period) with three workouts a week and a washout (no supplement) period of 2 weeks between supplementation periods. E is a combination of powder, containing protein and vitamin D, and capsules containing ω3 fatty acids. When on E, participants will receive 0.6 g protein/kg body weight, 20 μg vitamin D, and 1.8 g ω3 fatty acids daily. When on W, they will receive 0.6 g protein/kg body weight and, when on P, they will receive 0.6 g maltodextrin/kg body weight daily. The order of E, W, and P will be random and counterbalanced. Throughout the study, participants will be on isoenergetic nutritional plans to avoid differences in energy intake that might compromise the validity of the study. The dietary plans will be individualized and will provided 1.0 g protein/kg body weight/day.

Participants will undergo measurements of muscle strength, muscle endurance, aerobic capacity, and body composition prior to the first supplementation period, between periods, and after the third period. Also, blood amino acids, fatty acid acids, vitamin D, hematology, biochemistry, and hormones will be measured. To avoid bias, assessors will not know which supplement each participant is taking during each period.

The main hypotheses of the study are: 1) Consumption of E will increase lean body mass compared to W and P; 2) consumption of E will improve muscle strength, muscle endurance, and aerobic capacity compared to W and P; and 3) consumption of E will result in a better blood amino acid, fatty acid, and vitamin D profile.

ELIGIBILITY:
Inclusion Criteria:

* Regular training (mixed endurance and resistance training 3-6 times a week, 50 min each session, for the past 4-6 months) as assessed by gym records or questionnaires.
* Clearance from a pathologist or cardiologist to perform maximal exercise.
* Mixed isoenergetic diet for the past 4-6 months.

Exclusion Criteria:

* Smoking (even one cigarette or nicotine-containing device over the past 6 months).
* Any injuries to the musculoskeletal system that could interfere with the execution of training.
* Chronic disease.
* Fish or oyster allergy.
* Milk allergy.
* Pregnancy, lactation or planning a pregnancy within the duration of the study.
* Regular use of prescription medicine or supplements that might affect muscle function or recovery over the past month.
* Intermittent or religious fasting.
* Any vegetarian, ketogenic and protein diet.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid profile pre-supplementation | Within 2 days before the beginning of supplementation.
  Plasma amino acid profile (that is, the concentration of each individual amino acid) will be determined by liquid chromatography - mass spectrometry.
Plasma amino acid profile post-supplementation | Within 2 days after the end of supplementation.
  Plasma amino acid profile (that is, the concentration of each individual amino acid) will be determined by liquid chromatography - mass spectrometry.
Whole-blood fatty acid profile pre-supplementation | Within 2 days before the beginning of supplementation.
  Whole-blood fatty acid profile (that is, the concentration of each individual fatty acid) will be determined by gas chromatography.
Whole-blood fatty acid profile post-supplementation | Within 2 days after the end of supplementation.
  Whole-blood fatty acid profile (that is, the concentration of each individual fatty acid) will be determined by gas chromatography.
Maximal dynamic strength of shoulder muscles pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Maximal dynamic strength of shoulder muscles will be assessed by measurement of one-repetition maximum.
Maximal dynamic strength of shoulder muscles post-supplementation | Within 2 weeks after the end of supplementation.
  Maximal dynamic strength of shoulder muscles will be assessed by measurement of one-repetition maximum.
Force-velocity relationship of knee flexors and extensors pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Force-velocity relationship of knee flexors and extensors will be assessed in isokinetic dynamometer.
Force-velocity relationship of knee flexors and extensors post-supplementation | Within 2 weeks after the end of supplementation.
  Force-velocity relationship of knee flexors and extensors will be assessed in isokinetic dynamometer.
Aerobic fitness pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Aerobic fitness will be assessed by measurement of maximal oxygen uptake through a maximal graded exercise test on treadmill.
Aerobic fitness post-supplementation | Within 2 weeks after the end of supplementation.
  Aerobic fitness will be assessed by measurement of maximal oxygen uptake through a maximal graded exercise test on treadmill.
Lean and fat mass pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Lean and fat mass of the whole body and its parts (trunk, legs and arms) will be assessed by dual X-ray absorptiometry.
Lean and fat mass post-supplementation | Within 2 weeks after the end of supplementation.
  Lean and fat mass of the whole body and its parts (trunk, legs and arms) will be assessed by dual X-ray absorptiometry.

SECONDARY OUTCOMES:
Plasma vitamin D concentration pre-supplementation | Within 2 days before the beginning of supplementation.
  Vitamin D will be measured by liquid chromatography - mass spectrometry.
Plasma vitamin D concentration post-supplementation | Within 2 days after the end of supplementation.
  Vitamin D will be measured by liquid chromatography - mass spectrometry.
Muscle endurance pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Muscle endurance will be assessed by performing multiple sit-ups, knee flexions and knee extensions.
Muscle endurance post-supplementation | Within 2 weeks after the end of supplementation.
  Muscle endurance will be assessed by performing multiple sit-ups, knee flexions and knee extensions.
Force-velocity relationship of shoulder muscles pre-supplementation | Within 2 weeks before the beginning of supplementation.
  Force-velocity relationship of shoulder muscles will be assessed by a linear encoder.
Force-velocity relationship of shoulder muscles post-supplementation | Within 2 weeks after the end of supplementation.
  Force-velocity relationship of shoulder muscles will be assessed by a linear encoder.
Full blood count pre-supplementation | Within 2 days before the beginning of supplementation.
  Full blood count will be performed by flow cytometry.
Full blood count post-supplementation | Within 2 days after the end of supplementation.
  Full blood count will be performed by flow cytometry.
Biochemical analyses pre-supplementation | Within 2 days before the beginning of supplementation.
  Plasma glucose, triacylglycerols, total cholesterol, HDL cholesterol, LDL cholesterol, urea, and creatinine (all in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Biochemical analyses post-supplementation | Within 2 days after the end of supplementation.
  Plasma glucose, triacylglycerols, total cholesterol, HDL cholesterol, LDL cholesterol, urea, and creatinine (all in mg/dL) will be measured by chemiluminescence in an automated analyzer.
Plasma enzymes pre-supplementation | Within 2 days before the beginning of supplementation.
  Creatine kinase and γ-glutamyltransferase (both in U/L) will be measured by chemiluminescence in an automated analyzer.
Plasma enzymes post-supplementation | Within 2 days after the end of supplementation.
  Creatine kinase and γ-glutamyltransferase (both in U/L) will be measured by chemiluminescence in an automated analyzer.
Hormonal analyses pre-supplementation | Within 2 days before the beginning of supplementation.
  Plasma cortisol and testosterone (both in μg/dL) will be measured by immunoluminescence in an automated analyzer.
Hormonal analyses post-supplementation | Within 2 days after the end of supplementation.
  Plasma cortisol and testosterone (both in μg/dL) will be measured by immunoluminescence in an automated analyzer.
Internal load of exercise pre-supplementation | Within the first week of supplementation.
  The internal load of exercise will be assessed by telemetric heart rate sensors and software.
Internal load of exercise post-supplementation | Within the last week of supplementation (week 6).
  The internal load of exercise will be assessed by telemetric heart rate sensors and software.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Evaluation of Human Biological Performance, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided